CLINICAL TRIAL: NCT01885169
Title: Safety of Live-attenuated Influenza Vaccine (LAIV, Flumist®) in Patients With Cystic Fibrosis (CF)
Brief Title: LAIV (Flumist®) Administration in CF Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Ministere de la Sante et des Services Sociaux (Other); Canadian Cystic Fibrosis Foundation (Other); PHAC/CIHR Influenza Research Network (Other Government)
Responsible Party: Principal Investigator, Caroline Quach-Thanh, Pediatric Infectious Diseases, Medical Microbiologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2012-4621
Record Dates: First submitted 2013-06-20; First posted 2013-06-24 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Influenza; Vaccine
MeSH Terms: conditions — Cystic Fibrosis; Influenza, Human | interventions — FluMist

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — nasal swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cohort A: Participants with CF; Flumist®-naïve
  Interventions: Biological: Flumist®
- Cohort B: Siblings of Cohort A without CF; Flumist®-naïve
  Interventions: Biological: Flumist®
- Cohort C: Participants with CF; Flumist®-experienced
  Interventions: Biological: Flumist®

INTERVENTIONS:
Biological: Flumist® — The three cohorts will receive Flumist® and will be swabbed for inflammatory markers and viral shedding.
  Other Names: Live-attenuated influenza virus; LAIV

SUMMARY:
Influenza (the "flu") is one of the most common respiratory viruses associated with respiratory deteriorations in children and adolescents with cystic fibrosis. These deteriorations usually mean antibiotics, hospitalizations, and worsening of pulmonary function tests. A new flu vaccine has been recently approved for use in Canada (Flumist®). What is particular about this flu vaccine is that it is a spray in the nose, which mimics how influenza usually infects us. This particular vaccine protects children and adolescents much better than the regular injectable flu shot.

This new vaccine has been given to > 2,000 healthy children and to >2,000 children with asthma and well tolerated. The investigators want to know if Flumist® is well tolerated in children with CF and does not cause worsening of respiratory symptoms. The investigators will conduct a study where all participants will receive Flumist® in the nose. This study is particularly important because its results will provide safety information on a vaccine that is more efficacious for a population who needs safe and easy to administer protection against the flu.

DETAILED DESCRIPTION:
The literature demonstrates a significant impact of influenza on the disease course of children with cystic fibrosis (CF) and superior efficacy of live-attenuated influenza vaccine (LAIV - Flumist®) compared to trivalent inactivated vaccine (TIV) in healthy and asthmatic children and adolescents. LAIV has recently been approved for use in Canada in people aged 2-59 years. CF is described as a hyper-inflammatory disorder, with abnormal inflammatory signaling, excessive inflammatory response, and impairment in the resolution of inflammation that could be a risk for the development of adverse events after LAIV. Given the impact of influenza in CF patients, the likelihood of superior protection of LAIV, the hyper-inflammatory status of CF patients that could increase the risk of adverse events, and the scarcity of data on the safety of LAIV use in this population, the assessment of LAIV's safety profile in CF patients is necessary to determine whether the anticipated benefits associated with LAIV use will outweigh potential risks, mainly respiratory deterioration. Our study specifically aims to:

Aim 1: Explore the mucosal inflammatory response in participants exposed to LAIV: Using self-procured nasal swabs in 75 participants with CF (30 previously vaccinated and 45 LAIV naïve) and 45 healthy siblings, the investigators aim to explore: (a) the inflammatory response profiles in patients with and without CF before and after LAIV and (b) if participants' inflammatory profiles differ whether they report respiratory deteriorations after LAIV or not. As viral infections were shown to induce cytokines production (IL-1b IL-6, TNFa and CXCL-8 [IL-8]) in nasal secretions, the expression of these 4 inflammatory markers will be profiled using a multiplex cytokine detection kit after LAIV in participants with and without CF. The inflammatory signatures will be compared in patients with/without CF and with/without respiratory deteriorations.

Aim 2: Determine LAIV efficacy in preventing shedding of viral strains upon challenge: Using the same 75 participants with CF and 45 healthy siblings from aim 1, the investigators will compare the proportion of children shedding vaccine strains among the LAIV naïve and LAIV experienced. The clinical efficacy will be extrapolated from the efficacy in preventing shedding and derived as 1 - (% shedding in LAIV experienced/% shedding in LAIV naïve).

Aim 3: Assess LAIV safety in patients with CF: Compare the incidence of severe AEFI following LAIV in children with CF vaccinated with LAIV during the previous season (n = 70) compared to those without prior vaccination with LAIV (n = 45). Using a self-controlled case-series design, the investigators will compare the incidence of AEFI during the at-risk period (Day 1-28 post LAIV) and non at-risk period (Days 29-56). These incidence rate ratios will be compared in children with CF who are LAIV experienced and LAIV naïve.

Methods: The cohort of children with CF will be vaccinated with LAIV and followed for 56 days by phone for the development of severe adverse events following immunization (AEFI). Both periods (4 weeks) will be monitored using the same methodology: a diary for monitoring of symptoms and hospital charts. The cohort of children without CF will be vaccinated with LAIV and followed for 8 days by phone (one phone call on day 8) for the development of severe AEFIs.

A subgroup of participants with CF (30 LAIV experienced at MCH and 45 LAIV naïve in BC) and 45 participants without CF will be recruited to also provide self-procured nasal swabs on day 0 (before LAIV), and then on days 1,2, 4, and 7 for inflammatory markers and viral shedding.

Knowledge gained from this project will be used to determine LAIV safety in children with CF, a patient population in whom influenza has major health impacts and who could greatly benefit from a recommendation for LAIV preferential use. Moreover, the intranasal route of administration should make this vaccine more acceptable to patients that need yearly vaccination, thereby potentially increasing vaccination coverage. Patients with CF are also the population in whom the risk of adverse events with LAIV is the highest, given their baseline respiratory condition and inflammatory dysregulation. Therefore, if LAIV is well tolerated in this population, the investigators could generalize LAIV preferential use to other pediatric populations with chronic conditions.

ELIGIBILITY:
Inclusion Criteria:

* followed in one of the participating clinics
* considered in stable condition prior to enrollment as per their physician,

Exclusion Criteria:

* allergic to eggs or other vaccine components
* patients for whom LAIV is contraindicated (i.e. on oral steroids for an acute asthma exacerbation or with a medically-attended wheezing episode in the 7 days prior to immunization)
* participants with clinically significant nasal polyps
* have a significant febrile illness (oral temperature ≥ 380C) at day of vaccination
* pregnant women
* immunosuppressed subjects

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric patients with CF followed in clinics in the provinces of Quebec and British Columbia
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Risk of severe respiratory deterioration in the 28-day period after LAIV leading to unscheduled clinical visit or emergency department visit with or without a hospitalization, compared to the second 28-day period (D29-56). | at-risk period (Days 1-28 post LAIV) and non at-risk period (Days 29-56)

SECONDARY OUTCOMES:
Efficacy in preventing viral shedding | Days 1, 2, 4, and 7 after LAIV
  We will compare viral shedding in children with CF who are LAIV naïve vs. LAIV experienced. To follow viral shedding, 90 LAIV naïve participants with and without CF and 30 LAIV experienced participants with CF will provide self-procured nasal swabs on days 1, 2, 4, and 7 after LAIV.

OTHER OUTCOMES:
Inflammatory response in CFs in response to LAIV | Before LAIV (day 0), and days 1, 2, 4, and 7
  Viral infections were shown to induce the production of cytokines IL-1beta, IL-6, TNFalpha and CXCL-8 (IL-8) in nasal secretions. The expression of the 4 inflammatory markers will be profiled using a multiplex cytokine detection kit in CF participants after LAIV.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Quach-Thanh, MD, MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Caroline Quach-Thanh, MD, MSc, Study Director — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (3):
- Canada (3):
  - Vaccine Evaluation Centre, Vancouver, British Columbia
  - The Montreal Children's Hospital, Montreal, Quebec
  - Centre Hospitalier de l'Université Laval, Québec, Quebec